CLINICAL TRIAL: NCT04567732
Title: Randomized Double Blind Clinical Study on the Treatment of Bilateral Knee Arthrosis: Intra-articular Injection of Filtered Autologous Adipose Tissue Versus Placebo
Brief Title: Bilateral Knee Osteoarthritis: Intra-articular Injection of Filtered Autologous Adipose Tissue Versus Placebo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AdipoBil
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Bilateral Knee Osteoarthritis; Autologous Adipose Tissue
Keywords: Arthrosis; Osteoarthrosis; Degenerative joint disease; Knee degenerative joint disease.; Bilateral; Fat tissue
MeSH Terms: conditions — Osteoarthritis; Joint Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filtered Autologous Adipose Tissue (Experimental): based on randomization one of the two knees will be treated with a single injection of Filtered Autologous Adipose Tissue
  Interventions: Combination Product: injection of Filtered Autologous Adipose Tissue
- Placebo (Placebo Comparator): based on randomization one of the two knees will be treated with a single injection of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: injection of Filtered Autologous Adipose Tissue — Single injection of Filtered Autologous Adipose Tissue
  Arms: Filtered Autologous Adipose Tissue
Drug: Placebo — Single injection of Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the radiological and clinical outcomes comparing two different treatments (Filtered Autologous Adipose Tissue versus Placebo) in patients affecting bilateral knee osteoarthritis.

After be randomized, every patient will be treated in both legs, one leg with Adipose Tissue and the other one with Placebo.

DETAILED DESCRIPTION:
All patients who meet the inclusion criteria and giving written informed consent will be randomized.

Every patient will be treated with a single injection of Filtered Autologous Adipose Tissue in one knee and single injection of Placebo in the other, based on the randomization.

After the treatment patients will be followed up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. bilateral degenerative chondropathy of the knees showing at least a grade 2-3 kellgren-lawrence classification (absence of severe osteoarthritis)
2. An overall Pain subscale score of the Western Ontario and McMaster Universities Osteoarthritis Index between a value of 9 and 19.
3. Failure, intended as the persistence of symptomatology, after at least one conservative treatment cycle (pharmacological, physiotherapeutic or infiltrative treatment);
4. Ability and informed consent of patients to actively participate in the rehabilitation protocol and clinical and radiological follow-up;

Exclusion Criteria:

1. Patients incapable of understanding and wanting;
2. Diagnosis of leukaemia, known presence of metastatic malignant cells, ongoing or planned chemotherapy;
3. Diagnosis of rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis or arthritis resulting from another inflammatory disease; infection with human immunodeficiency virus (HIV), viral hepatitis; chondrocalcinosis;
4. Patients with uncontrolled diabetes mellitus;
5. Patients with uncontrolled thyroid metabolic disorders;
6. Patients who abuse alcoholic beverages, drugs or medicines;
7. Patients with misalignment of the lower limbs above 10 degrees;
8. Body Mass Index > 40;
9. Pregnant or lactating state or intention to become pregnant during the period of participation in the study.
10. Patients with a history of trauma or intra-articular infiltration of therapeutic substances in the 6 months prior to screening.
11. Patients who have had knee surgery in the 12 months prior to screening.
12. Patients with insufficient abdominal adipose tissue, assessed by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 months
  It is a 0 - 100 standardized questionnaire widely used for the evaluation of patients with knee osteoarthrosis. The questionnaire is made by three subscale: Pain (5 questions ranging from 0 - 20), Stiffness (2 questions ranging from 0 - 8) and Function (17 questions ranging from 0 - 68).

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 1, 3, 6, and 24 months
  It is a 0 - 100 standardized questionnaire widely used for the evaluation of patients with knee osteoarthrosis. The questionnaire is made by three subscale: Pain (5 questions ranging from 0 - 20), Stiffness (2 questions ranging from 0 - 8) and Function (17 questions ranging from 0 - 68).
Subjective International Knee Documentation Committee (IKDC - subjective score) | Baseline, 1, 3, 6, 12 and 24 months
  Questionnaire is specific for knee pathologies. it is composed by three subscales: Symptoms, Sport Activities and Knee Function. (Total score 0-100)
Objective International Knee Documentation Committee (IKDC-Objective Score) | Baseline, 1, 3, 6, 12 and 24 months
  The presence of effusions and the degree of movement of the knee are evaluated, the worst value of one of these parameters determines the final value of the IKDC degree. There are four grades (A, B, C, D) which respectively identify a knee rated as normal, near normal, abnormal and severely abnormal;
Tegner score | Before symptoms onset, at the baseline
  describe and assess the sport activity with a score ranging from 0 to 10, where 0 means "inability" and 10 represent ability to perform "competitive sports".
Patient Acceptable Symptom State (PASS) | Baseline, 1, 3, 6, 12 and 24 months
  tool for assessing patient satisfaction in consideration of their current degree of pain, function and daily activity. The patient will evaluate his degree of satisfaction by answering a dichotomous closed question (yes / no).
EuroQol Visual Analogue Scale (EQ-VAS) | Baseline, 1, 3, 6, 12 and 24 months
  0 - 100 scale where 100 is the "best possible health"and 0 is the "worst possible health"
Numeric Rating Scale (NRS) - Function | Baseline, 1, 3, 6, 12 and 24 months
  the scale is to expect the patient to select the number that best describes their functional disability status, from 0 to 10. The higher the value indicated the higher the degree of disability will be.
Numeric Rating Scale (NRS) - Pain | Baseline, 1, 3, 6, 12 and 24 months
  the scale requires the patient to select the number that best describes the intensity of his pain, from 0 to 10, at that precise moment. 0 means no pain and 10 means worst possible pain.
Kellgren-Lawrence score | baseline and 24 months
  grade 0 to 4 for the assessment of the knee osteoarthritis grade, where 4 is the worst possible grade.
Magnetic Resonance Imaging | baseline and 12 months
  evaluation of the knee joint
overall judgement on the treatment | 6, 12 and 24 months
  The patient must indicate the degree of satisfaction with the treatment carried out at the end of the clinical trial

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Bianchi F, Maioli M, Leonardi E, Olivi E, Pasquinelli G, Valente S, Mendez AJ, Ricordi C, Raffaini M, Tremolada C, Ventura C. A new nonenzymatic method and device to obtain a fat tissue derivative highly enriched in pericyte-like elements by mild mechanical forces from human lipoaspirates. Cell Transplant. 2013;22(11):2063-77. doi: 10.3727/096368912X657855. Epub 2012 Oct 8. PMID 23051701
- [Background] Tremolada C, Palmieri G, Ricordi C. Adipocyte transplantation and stem cells: plastic surgery meets regenerative medicine. Cell Transplant. 2010;19(10):1217-23. doi: 10.3727/096368910X507187. Epub 2010 May 4. PMID 20444320
- [Background] Perdisa F, Gostynska N, Roffi A, Filardo G, Marcacci M, Kon E. Adipose-Derived Mesenchymal Stem Cells for the Treatment of Articular Cartilage: A Systematic Review on Preclinical and Clinical Evidence. Stem Cells Int. 2015;2015:597652. doi: 10.1155/2015/597652. Epub 2015 Jul 9. PMID 26240572
- [Background] Koh YG, Kwon OR, Kim YS, Choi YJ. Comparative outcomes of open-wedge high tibial osteotomy with platelet-rich plasma alone or in combination with mesenchymal stem cell treatment: a prospective study. Arthroscopy. 2014 Nov;30(11):1453-60. doi: 10.1016/j.arthro.2014.05.036. Epub 2014 Aug 6. PMID 25108907
- [Background] Bellamy N, Hochberg M, Tubach F, Martin-Mola E, Awada H, Bombardier C, Hajjaj-Hassouni N, Logeart I, Matucci-Cerinic M, van de Laar M, van der Heijde D, Dougados M. Development of multinational definitions of minimal clinically important improvement and patient acceptable symptomatic state in osteoarthritis. Arthritis Care Res (Hoboken). 2015 Jul;67(7):972-80. doi: 10.1002/acr.22538. PMID 25581339